CLINICAL TRIAL: NCT03150342
Title: Presentations of Hypertrophic Cardiomyopathy on Myocardial Perfusion Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Szu-Ying Tsai, Resident Physician, department of nuclear medicine, Far Eastern Memorial Hospital
Other Study IDs: 106057-E
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Hypertrophic Cardiomyopathy; Myocardial Perfusion Imaging
Keywords: CZT scanner; myocardial perfusion imaging; Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Myocardial Perfusion Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: myocardial perfusion imaging — dipyridamole-stressed MPI scan using thallium-201

SUMMARY:
Chest pain and myocardial ischemia are prevailing features in patients with hypertrophic cardiomyopathy (HCM). Recently introduced single-photon emission computed tomography (SPECT) cameras with solid-state cadmium-zinc-telluride (CZT) detectors have been shown to decrease imaging time and improved the imaging quality of gated myocardial perfusion imaging (MPI). The investigators also correlate the MPI parameters with echocardiographic parameters. This study is to examine the spatial distribution of stress perfusion abnormalities and tissue injury in patients with HCM using a CZT SPECT camera.

DETAILED DESCRIPTION:
The investigators will retrospectively evaluate myocardial perfusion patterns and cardiac function with Thallium (Tl)-201 gated dipyridamole MPI in patients with clinical diagnosis of HCM and patent coronary angiography between January 2013 and October 2016. The inclusion criteria included a spade-like configuration on left ventriculogram, or echocardiographic findings suggestive of HCM. The participants will be then divided into the following three groups: apical, concentric and septal forms. Regional perfusion would be analyzed using a 17-segment model from 0-4 degree (0=normal, to 4=absent perfusion); and summed stress score (SSS), summed rest score (SRS) and summed difference score (SDS) were calculated. Gated SPECT would be processed by quantitative gated SPECT (QGS) software (Cedars-Sinai Medical Center, Los Angeles, CA, USA) and ejection fraction phase analysis. Diastolic parameters would be also acquired by Doppler echocardiography, and correlated with MPI parameters.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of HCM and patent coronary angiography between January 2013 and October 2016.

Exclusion Criteria:

* patient with prior myocardial ischemia, conduction abnormality, valvular disease or other cardiomyopathy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCM patients with patent coronary artery who underwent MPI
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-08-31 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
MPI results | January 2013 and October 2016.
  including perfusion abnormalities, and ejection fraction phase analysis results

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Wen Wu, MD, PhD, Study Director — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan